CLINICAL TRIAL: NCT04198753
Title: Skin Characteristics of Parents of Food Allergic Pediatric Patients
Status: Suspended | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3257
Record Dates: First submitted 2019-11-12; First posted 2019-12-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Food Allergy in Children
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parent of Peanut Allergic Child: The researchers will identify patients or study subjects aged 1-18 who have been diagnosed with peanut allergy based on skin prick testing, serologic testing, and/or history of reaction. They will then contact mothers or fathers of these patients/subjects who are 18 and older and enroll those who do not themselves have a history of food allergy, with a goal of 40 subjects per group.
  The researchers will perform a very limited physical exam followed by skin tape stripping (30 strips) for lipid profile and protein expression, and transepidermal water loss (TEWL) measurements every 5 strips. They will obtain blood work to define FLG mutation and vitamin D status. Questionnaires on their background, other concurrent atopic and nonatopic diseases, and exposures, will also be collected.
  Interventions: Diagnostic Test: Skin tape stripping; Device: Skin barrier assessment; Diagnostic Test: Blood draw
- Parent of Non-atopic Child: To establish normal controls, the researchers will enroll parents age 18 or older with no history of food allergy or eczema in themselves or their offspring.
  The researchers will perform a very limited physical exam followed by skin tape stripping (30 strips) for lipid profile and protein expression, and transepidermal water loss (TEWL) measurements every 5 strips. They will obtain blood work to define FLG mutation and vitamin D status. Questionnaires on their background, other concurrent atopic and nonatopic diseases, and exposures, will also be collected.
  Interventions: Diagnostic Test: Skin tape stripping; Device: Skin barrier assessment; Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Skin tape stripping — Adhesive skin sampling discs will be firmly pressed against the skin in a hairless location (not the face) followed by lifting it free of the skin. Tape stripping will be collected from non-lesional skin up to 30 times. These discs will then be used to evaluate proteins and lipids. With every 5 tape strips collected, transepidermal water loss measurements will be performed.
Device: Skin barrier assessment — A small device will be used to measure transepidermal water loss (TEWL), which is the quantity of water that passes from inside the body through the skin to the surrounding atmosphere via diffusion and evaporation process. The device, a probe, is simply placed against the skin surface making superficial contact and kept there for a few seconds until the measurement terminates. This will be performed at baseline and after every 5 tape strips.
Diagnostic Test: Blood draw — Subjects will undergo genetic testing of FLG mutation status (5mL of whole blood in lavender top tube) and vitamin D level (2mL of whole blood in red top tube) via blood draw.

SUMMARY:
The purpose of this study is to determine whether disruptions in the skin barrier of parents can contribute to the development of food allergies in their offspring. The study team will compare the superficial skin layers of mothers and fathers who do not have children with diagnosed food allergies to the skin layers of parents who do have children with diagnosed food allergy. The study will include a questionnaire, noninvasive superficial skin testing with skin tapping and transepidermal water loss measurements, and a blood draw.

DETAILED DESCRIPTION:
There is an already well-established link between atopic dermatitis (AD), or eczema, and the development of food allergies. More specifically, it is believed that sensitizations to food can occur through low-dose cutaneous sensitization via a disrupted skin barrier. The strongest genetic contributor to eczema is the FLG loss-of-function or missense mutation, which is associated with increased transepidermal water loss and increased skin permeability (1). In a recent study exploring the risk of maternal transmission of allergic risk, it was found that children of FLG-carrier mothers had a 1.5 increased AD risk, specifically when these mothers had allergic sensitization (elevated allergen-specific IgE antibody plasma levels) but independent of their own FLG mutation status (10). This information may suggest that an interrupted skin barrier in mothers may serve as an environmental risk factor for the development of food allergies in their offspring.

The purpose of our study is to evaluate the skin characteristics and FLG gene mutation status of parents of known food allergic pediatric patients. The researchers hypothesize that parents of food allergic patients will have more significant disruptions in their skin barrier function than parents of children who do not suffer from food allergies.

In order to evaluate skin barrier disruptions in these subjects, two noninvasive methods will be performed including skin tape stripping, a total of 30 strips per subject, and transepidermal water loss measurements using a small device. Both methods are relatively painless and cause minimal risk to the participant. In order to evaluated FLG gene mutation status, blood draw will also be performed. Subjects will undergo a focused physical exam and also be requested to fill out a detailed questionnaire. The researchers will obtain additional offspring peanut allergy clinical characteristics from the medical records. All data collection will occur over 1-2 visits, averaging an anticipated 1 hour in total duration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the informed consent form
2. 18 years of age or older (inclusive) 3. One of the following Diagnostic Categories:

   1. Normal healthy controls with no personal or offspring history of food allergy or atopic dermatitis
   2. Mother or father without personal history of food allergy, but with a child diagnosed with peanut allergy. Peanut allergy is defined as fulfilling one of the following 3 criteria:

   i. Clinical history defined as one of the following occurring within 2 hours of exposure to peanut:
   1. Involvement of the skin-mucosal tissue (eg, generalized hives, itch-flush, swollen lips-tongue-uvula)
   2. Respiratory compromise (eg, dyspnea, wheeze-bronchospasm, stridor, reduced PEF, hypoxemia)
   3. Reduced BP or associated symptoms (eg, hypotonia [collapse], syncope, incontinence)
   4. Persistent gastrointestinal symptoms (eg, crampy abdominal pain, vomiting)

ii. Positive skin prick testing > 8 mm

iii. Positive specific IgE to peanut > 14.0 kUA/L

Exclusion Criteria:

1. Has active flare of atopic dermatitis requiring use of bleach baths, topical corticosteroids, topical immunomodulatory agents, or topical antibiotics on the extremity being evaluated
2. Has a skin disease other than AD that might compromise the stratum corneum barrier such as bullous disease, psoriasis, cutaneous T cell lymphoma, Darier's disease, HaileyHailey, or dermatitis herpetiformis
3. Has a current systemic infection requiring use of systemic antibiotics, antiparasitics, antivirals, or antifungals
4. Has a severe concomitant disease or immunosuppression such as lymphoma, HIV, or Wiskott-Aldrich syndrome
5. Has a history of a severe reaction to latex, tape, or adhesives
6. Has used any biologics within 5 half-lives or 16 weeks, whichever is longer
7. Has received immunotherapy in the last 12 months
8. Has used any investigational drugs within 5 half-lives or 8 weeks, whichever is longer
9. Has used anticoagulants, anxiolytics, or antidepressants within 30 days
10. Has used of systemic immunosuppressive drugs including oral steroids within 30 days
11. Has received total body phototherapy (e.g., ultraviolet light B [UVB], psoralen plus ultraviolet light A [PUVA], tanning beds [>1 visit per week]) within 30 days
12. Is pregnant or lactating (this will be self-verified by the patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Peanut allergic patients/subjects will be identified via the NJH EMR or database. Parents may be approached by listed study staff at the beginning or end of their scheduled NJH visit and asked about their food allergy history and interest in enrollment. Alternatively, this may be done over the phone. Thereafter, eligibility will be determined using the listed inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-06 (Estimated)

PRIMARY OUTCOMES:
Skin barrier dysfunction via skin tape stripping (STS) | 6-12 months
  To determine the level of skin barrier dysfunction in parents of peanut allergic (PA) patients versus parents of nonatopic (no food allergies, atopic dermatitis, or allergic rhinitis) patients using tape stripping.
Skin barrier dysfunction via transepidermal water loss (TEWL) measurements | 6-12 months
  To determine the level of skin barrier dysfunction in parents of peanut allergic (PA) patients versus parents of nonatopic (no food allergies, atopic dermatitis, or allergic rhinitis) patients using TEWL assessments.

SECONDARY OUTCOMES:
FLG mutation status | 6-12 months
  To determine filaggrin gene mutation status and evaluate if this correlates to the level of skin barrier dysfunction found on skin tape stripping and TEWL assessments.
Vitamin D status | 6-12 months
  To determine vitamin D status and evaluate if this correlates to the level of skin barrier dysfunction found on skin tape stripping and TEWL assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lack G. Update on risk factors for food allergy. J Allergy Clin Immunol. 2012 May;129(5):1187-97. doi: 10.1016/j.jaci.2012.02.036. Epub 2012 Mar 30. PMID 22464642
- [Background] Esparza-Gordillo J, Matanovic A, Marenholz I, Bauerfeind A, Rohde K, Nemat K, Lee-Kirsch MA, Nordenskjold M, Winge MC, Keil T, Kruger R, Lau S, Beyer K, Kalb B, Niggemann B, Hubner N, Cordell HJ, Bradley M, Lee YA. Maternal filaggrin mutations increase the risk of atopic dermatitis in children: an effect independent of mutation inheritance. PLoS Genet. 2015 Mar 10;11(3):e1005076. doi: 10.1371/journal.pgen.1005076. eCollection 2015 Mar. PMID 25757221
- [Background] Broccardo CJ, Mahaffey SB, Strand M, Reisdorph NA, Leung DY. Peeling off the layers: skin taping and a novel proteomics approach to study atopic dermatitis. J Allergy Clin Immunol. 2009 Nov;124(5):1113-5.e1-11. doi: 10.1016/j.jaci.2009.07.057. Epub 2009 Sep 12. No abstract available. PMID 19748658
- [Background] Kelleher M, Dunn-Galvin A, Hourihane JO, Murray D, Campbell LE, McLean WHI, Irvine AD. Skin barrier dysfunction measured by transepidermal water loss at 2 days and 2 months predates and predicts atopic dermatitis at 1 year. J Allergy Clin Immunol. 2015 Apr;135(4):930-935.e1. doi: 10.1016/j.jaci.2014.12.013. Epub 2015 Jan 22. PMID 25618747 (Retraction: PMID 33832697 J Allergy Clin Immunol. 2021 Apr;147(4):1526)